CLINICAL TRIAL: NCT04961229
Title: Booster Dose of mRNA SARS-CoV-2 Vaccine for Kidney Transplant Recipients Without Adequate Humoral Response With or Without Immunosuppression Reduction - Protocol for a Randomised Controlled Trial (BECAME Study)
Brief Title: Booster Dose of COVID-19 Vaccine for Kidney Transplant Recipients Without Adequate Humoral Response
Acronym: WHO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: dafna yahav (Other)
Responsible Party: Sponsor-Investigator, dafna yahav, Clinical Professor, Infectious Diseases Unit, Rabin Medical Center, Beilinson Campus, Petah-Tikva, Israel, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0192-21-RMC
Record Dates: First submitted 2021-07-13; First posted 2021-07-14 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Immunosuppression
Keywords: kidney transplant recipients; COVID-19; vaccine; immunosuppression reduction; randomized controlled trial
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Third dose of BNT162b2 vaccine with Immunosuppression reduction (Experimental): Third dose of BNT162b2 vaccine with reduction of mycophenolic acid dose
  Interventions: Biological: The Pfizer mRNA-based BNT162b2 vaccine
- Third dose of BNT162b2 vaccine without immunosuppression reduction (Experimental): Third dose of BNT162b2 vaccine without reduction of mycophenolic acid dose
  Interventions: Biological: The Pfizer mRNA-based BNT162b2 vaccine
- Third dose of BNT162b2 vaccine (Experimental): Third dose of BNT162b2 vaccine with no change in immunosuppression for patients that are excluded from the randomised trial
  Interventions: Biological: The Pfizer mRNA-based BNT162b2 vaccine

INTERVENTIONS:
Biological: The Pfizer mRNA-based BNT162b2 vaccine — participants who gave informed consent to participate in either the prospective non-randomised study or RCT will receive a single vaccine dose.
  In addition, participants in the RCT will be randomised into two groups:
  1. Third booster dose of BNT162b2 (one standard dose) with no change in immunosuppression protocol
  2. Third booster dose of BNT162b2 (one standard dose) with immunosuppression reduction according to protocol (mycophenolic temporary cessation 4 days before (5 half-lives) and one week (expected antibody response) after vaccination (to allow for antibody response).

SUMMARY:
Introduction: Inadequate antibody response to mRNA SARS-CoV-2 vaccination has been described among kidney transplant recipients. Immunosuppression level and specifically, use of antimetabolite in the maintenance immunosuppressive regimen, are associated with inadequate response. In light of the severe consequences of COVID-19 in solid organ transplant recipients, we believe it is justified to examine new vaccination strategies in these patients.

Methods and analysis: BECAME is a single center, open label, investigator-initiated randomised controlled, superiority trial, aiming to compare immunosuppression reduction combined with a third BNT162b2 vaccine dose versus third dose alone. The primary outcome will be seropositivity rate against SARS-CoV-2. A sample size of 154 patients was calculated for the seropositivity endpoint assuming 25% seropositivity in the control group and 50% in the intervention group. A sample of participant per arm will be also teste for T-cell response. We also plan to perform a prospective observational study, evaluating seropositivity among ~350 kidney transplant recipients consenting to receive a third vaccine dose, who are not eligible for the randomised controlled trial.

Ethics and dissemination: The trial is approved by local ethics committee of Rabin medical center (RMC-0192- 21). Results of this trial will be published; trial data will be available. Protocol amendments will be submitted to the local ethics committee.

DETAILED DESCRIPTION:
All recipients more than 6 months post transplantation and at least 3 weeks following second vaccine dose will be approached and invited to a first study visit.

At first visit:

* Signed informed consent will be obtained from participants willing to participate by study investigators who usually work in the transplantation clinic.
* Anti-spike antibody response will be assessed using SARS-CoV-2 IgG II Quant (Abbott©) assay. Participants who have a documented seronegative test in the last 6 weeks will not be tested again.

Participants will be invited for an additional visit once negative serology will be reported, within 7 days of serology collection. At this second visit all participants who gave informed consent to participate in either the prospective non-randomised study or RCT will receive a single vaccine dose.

In addition, participants in the RCT will be randomised into two groups:

1. Third booster dose of BNT162b2 (one standard dose) with no change in immunosuppression protocol
2. Third booster dose of BNT162b2 (one standard dose) with immunosuppression reduction according to protocol (mycophenolic temporary cessation 4 days before (5 half-lives) and one week (expected antibody response) after vaccination (to allow for antibody response).

Patients who will test seronegative will be informed by the study coordinator by phone in which study arm they will be participating and receive instructions for immunosuppression reduction both during the phone call and by written instructions provided to each patient during the first visit (see Appendix). Participants in the observational study will receive a third vaccine standard dose, without any change in immunosuppression (beyond routine care)

For all groups:

* Antibodies titer against spike protein will be evaluated again 2 weeks and 3, 6, 12 months after the third vaccine dose
* T-cell response will be evaluated for a subset of patients in each group (estimated 20 patients per arm) before booster dose, at 2 weeks after booster dose, and at 3 months. For T cell response quantification peripheral blood mononuclear cell (PBMC) will be stimulated for 24 hours with spike protein and secreted interferon-gamma (IFNg) will be measured by ELISA.
* Follow-up for adverse events, rejection and SARS-CoV-2 infection will be performed at 2 weeks and at three, 6 and 12 months post third vaccination dose

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant recipients that received two doses of BNT162b2 vaccine at least 3 weeks prior to enrollment, and were seronegative (IgG against the spike protein of SARS-CoV-2 below 50 AU/ml) at least two weeks after the second vaccine dose

Additional inclusion criteria for the RCT:

* Recipients treated by three anti-rejection medications including: prednisone, tacrolimus, mycophenolate mofetil or mycophenolic acid.
* Tacrolimus trough blood levels 5-10 nGr/ml (lower or higher doses will have to be adjusted before re-considering for inclusion)

Exclusion Criteria:

* Past infection with SARS-CoV-2
* Pregnancy
* Age below 18 years
* Active infection

Additional exclusion criteria for RCT only:

- Recipients at a high risk for acute or chronic humoral rejection including:

* Recipients with positive panel-reactive antibody (PRA) (any positive value) at any time before or after transplantation
* Recipients that had an acute rejection in the last year
* Recipients less than 6 months after transplantation
* Recipients that are considered at high risk for rejection according to the primary care nephrologist
* Recipients taking less than 3 anti-rejection medications
* Recipients currently treated with mTOR inhibitors (everolimus, sirolimus) and/or azathioprine
* Recipients treated with plasmapheresis in the previous 3 months
* Recipients treated with eculizumab in the last year
* Recipient treated with IVIG in the previous 3 months
* Recipient treated with rituximab in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
anti-spike protein titer above 50 AU/ml 2 weeks post vaccination | 2 weeks post vaccination
  positive humoral response against SARS-CoV-2

SECONDARY OUTCOMES:
anti-spike protein titer above 50 AU/ml 3-, 6-, and 12-months post vaccination | 3-, 6-, and 12-months post vaccination
  positive humoral response against SARS-CoV-2
Log transformed titer of anti-spike protein weeks and 3, 6, and 12 months post vaccination | 2 weeks and 3, 6, and 12 months post vaccination
  Log transformed titer of anti-spike protein
Adverse events to booster dose using CTCAE v4.0 criteria | 2 weeks post vaccine
  Severity of adverse events will be assessed using CTCAE v4.0 criteria
Acute rejection of the allograft either documented by biopsy or clinically suspected, defined as increase in creatinine by 20% from baseline, without any other plausible explanation | 2 weeks, 3,6, and 12 months post vaccination
  either documented by biopsy or clinically suspected, defined as increase in creatinine by 20% from baseline, without any other plausible explanation
positive PCR test to SARS-CoV-2 during the follow up period | until 12 months following vaccine
  positive PCR test to SARS-CoV-2 during the follow up period
Positive PCR tests to VZV, CMV | during the follow up period
  Other viral reactivation during the follow up period: VZV, CMV, tested according to clinical suspicion
Number of hospitalizations (numerical count) | until 12 months following vaccine
  Number of hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Rahaminov, Principal Investigator — Rabin Medical Center, Beilinson Campus, Petah-Tikva, Israel

IPD SHARING:
Plan to Share IPD: Yes
According to request
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available once entered for all patients and analyzed, presumably at 1-January-2022. It will be available for one year.
Access Criteria: Researchers who would like to share the data will be requested to send the PI their protocol/reason for asking the data. After reviewing the request, if the protocol seems adequate in terms of clinical question and methodological quality, we will share anonymized data.

REFERENCES:
- [Derived] Yahav D, Rozen-Zvi B, Mashraki T, Atamna A, Ben-Zvi H, Bar-Haim E, Rahamimov R. Immunosuppression reduction when administering a booster dose of the BNT162b2 mRNA SARS-CoV-2 vaccine in kidney transplant recipients without adequate humoral response following two vaccine doses: protocol for a randomised controlled trial (BECAME study). BMJ Open. 2021 Oct 11;11(10):e055611. doi: 10.1136/bmjopen-2021-055611. PMID 34635537